CLINICAL TRIAL: NCT01141894
Title: Evaluation of Costs and Consequences of Alternative Strategies of Intraoperative Fluid and Pharmacological Optimization. A Randomized Clinical Trial
Brief Title: Goal Directed Haemodynamic Treatment for Patients With Proximal Femoral Fracture
Acronym: GDHT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erzsebet Bartha, Medical Doctor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-018087-10; ID: 2008-1240-31 (Other: Ethical Board of Karolinska Institute Stockholm)
Record Dates: First submitted 2010-04-20; First posted 2010-06-11 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Femoral Fracture
Keywords: Proximal Femoral Fracture
MeSH Terms: conditions — Femoral Fractures; Proximal Femoral Fractures | interventions — Dobutamine; HES 130-0.4; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine fluid treatment (Active Comparator): Buffered Glucose 25 mg/ml 1ml/kg/h Ringer's Acetate 2 ml/kg/h and additionally as needed Voluven at the attending anaesthetist's discretion Phenylephrine 50 μg for correction of hypotension
  Interventions: Other: Routine fluid treatment
- Goal directed haemodynamic treatment (Experimental): Goal directed haemodynamic treatment Dobutamine 0.2-10 μg/kg/min Buffered Glucose 25 mg/ml 1ml/kg/h Ringer's Acetate 2 ml/kg/h Voluven 3 ml/kg as fluid challenge at the attending anaesthetist's discretion Phenylephrine 50 μg for correction of hypotension
  Interventions: Other: Goal directed haemodynamic treatment

INTERVENTIONS:
Other: Goal directed haemodynamic treatment — Treatment by fluids and Dobutamine to attain fixed haemodynamic goal
  Other Names: Dobutamine 0.2-10 μg/kg/min; Buffered Glucose 25 mg/ml 1 ml/kg/h; Ringer´s Acetate 2 ml/kg/h; Voluven 3 ml/kg as fluid challenge; Phenylephrine 50 μg for correction of hypotension
  Arms: Goal directed haemodynamic treatment
Other: Routine fluid treatment — Protocol guided fluid treatment used in the clinical routine
  Other Names: Buffered Glucose 25 mg/ml 1ml/kg/h; Ringer´s Acetate 2 ml/kg/h; Voluven at the attending anaesthetist's discretion; Phenylephrine 50 μg for correction of hypotension
  Arms: Routine fluid treatment

SUMMARY:
The investigators aimed to compare the costs and consequences of 'routine perioperative fluid therapy' and 'GDHT in terms of morbidity, mortality, length of hospital stay, activity of daily living, health related quality of life, cognitive functions and need of social services and up till 12 months following operations of proximal femoral fracture at elderly. The primary hypothesis is that 'GDHT is a better strategy than 'routine fluid therapy' in terms of reduced frequency of postoperative complications.

DETAILED DESCRIPTION:
The investigation is an open, randomized clinical study of individuals suffering from a proximal femoral fracture. The total study duration for each subject is approximately 12 months (+- 1 month); each patient will have 4'visits' (i.e. when PI extracts data to database) including regular praxis total: at registration; at discharge; 4 months and finally at 12 months after the surgery. For practical and logistic reasons, an interim-analysis will be conducted after approximately 100 patients whose data are completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients (men and women) age ≥ 70 years
* Patients´ scheduled for operation of proximal femoral fracture during office hours
* Patient who have a witnessed or written informed consent

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

* Concomitant medication with Lithium
* Known allergy (or hypersensitivity) to Lithium, or components of the medical device
* Weight ≤ 40 kg
* Other conditions or symptoms preventing the subject from entering the study, according to investigators judgment
* Life expectancy less than 6 months and/or pathological fractures
* Not possible to insert arterial line.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
number of patients with postoperative complications | up to 2 weeks
  absolute value, number

SECONDARY OUTCOMES:
Health Related Quality of Life | 1 year
  European Quality of Life questionaire using five dimensions (EQ-5D)shall be registered preoperatively, at 4 and 12 months postoperatively
number of complications | 4 months
  absolute value number
number of complications | 12 months
  absolute value number
health related quality of life | 4 months
health related quality of life | 12 months
  absolute value number
haemodynamic parameters | baseline
  monitor readings from LiDCO plus

CONTACTS AND LOCATIONS:
Overall Officials: Erzsebet Bartha, M.D, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Sweden

REFERENCES:
- [Derived] Bartha E, Arfwedson C, Imnell A, Kalman S. Towards individualized perioperative, goal-directed haemodynamic algorithms for patients of advanced age: observations during a randomized controlled trial (NCT01141894). Br J Anaesth. 2016 Apr;116(4):486-92. doi: 10.1093/bja/aew025. PMID 26994228
- [Derived] Bartha E, Davidson T, Brodtkorb TH, Carlsson P, Kalman S. Value of information: interim analysis of a randomized, controlled trial of goal-directed hemodynamic treatment for aged patients. Trials. 2013 Jul 9;14:205. doi: 10.1186/1745-6215-14-205. PMID 23837606